CLINICAL TRIAL: NCT00897338
Title: A Feasibility Study of a Novel Technique to Identify Circulating Breast Cancer Cells in Patients With Metastatic Breast Cancer
Brief Title: Identifying Circulating Breast Cancer Cells in Women With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0737 CDR0000571962; P30CA006973 (NIH); JHOC-J0737
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Flow Cytometry; Immunohistochemistry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: flow cytometry — laboratory analysis
Other: fluorescence activated cell sorting — laboratory analysis
Other: immunohistochemistry staining method — laboratory analysis
Other: immunologic technique — laboratory analysis
Other: biomarker analysis — laboratory analysis

SUMMARY:
RATIONALE: Studying samples of blood and pleural or peritoneal fluid from patients with metastatic breast cancer in the laboratory may help doctors identify biomarkers related to breast cancer and learn more about how breast cancer begins and spreads in the body.

PURPOSE: This research study is looking at a new way of identifying circulating breast cancer cells in blood and in pleural or peritoneal fluid in women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare identification of circulating breast cancer cells (CBCCs) in blood or pleural or peritoneal fluid by a novel technique using stem cell marker retinaldehyde dehydrogenase (ALDH) and surface antigen expression (CD44+, CD24-) to the standard technique using the CellSearch® system in women with metastatic breast cancer.

Secondary

* To determine whether CBCCs have the potential to grow into metastatic lesions.

OUTLINE: Patients undergo sample collection to help develop a new technique using stem cell marker retinaldehyde dehydrogenase (ALDH) and surface antigen expression (CD44+, CD24-) in isolating circulating breast cancer cells (CBCCs) from blood and pleural or peritoneal fluid. Blood may also be drawn to measure the number of circulating tumor cells using the standard CellSearch® system.

Mononuclear cells are isolated by density centrifugation. Cells are stained against surface antigens that provide specific expression patterns for CBCCs (CD44, CD24). Cells are analyzed on a fluorescence activated cell sorting (FACS) Calibur flow cytometer and sequentially gated (ALDHhigh→CD44+ vs CD24-/low or CD44+ vs CD24-/low→ALDHhigh) for detection of CBCCs. For further confirmation of epithelial origin, ALDHhighCD44+CD24-/low cells are isolated using a FACSAria flow sorter, cytocentrifuged onto glass slides then stained for the expression of epithelial-specific cytokeratins 5, 8, 14, 18 and 19 by standard immunohistochemical techniques. Using the phenotype that is found to most highly enrich for epithelial cells, cells are isolated by FACS and assayed for clonogenic growth.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Metastatic disease (stage IV)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic breast cancer patients
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2007-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of novel technique to identify and isolate circulating breast cancer cells | Baseline
Comparison of this novel technique with the CellSearch™ system | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States